CLINICAL TRIAL: NCT01473069
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety,Tolerability and Pharmacokinetics of Multiple Ascending Doses of JTK-853 Administered for Two Weeks in Healthy Subjects
Brief Title: Two Week Study Evaluating Safety, Tolerability and Pharmacokinetics of Multiple Doses of JTK-853 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK853-U-10-003
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: JTK-853; Healthy subjects
MeSH Terms: interventions — JTK-853; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose 1 JTK-853, 400 mg ketoconazole (Experimental)
  Interventions: Drug: JTK-853, ketoconazole
- Dose 2 JTK-853 (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 3 JTK-853 (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Dose 4 JTK-853 (Experimental)
  Interventions: Drug: JTK-853 or Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: JTK-853 or Placebo

INTERVENTIONS:
Drug: JTK-853, ketoconazole — JTK-853 Tablets or Placebo, twice a day for 14 days, JTK-853 and ketoconazole Tablets, 1 each on Day 15
  Arms: Dose 1 JTK-853, 400 mg ketoconazole
Drug: JTK-853 or Placebo — JTK-853 Tablets or Placebo, twice a day for 14 days
  Arms: Dose 2 JTK-853; Dose 3 JTK-853; Dose 4 JTK-853; Placebo

SUMMARY:
The purpose of this study was to determine the safety, tolerability and pharmacokinetics of sequential ascending doses of JTK-853 administered for 14 days in healthy subjects and also to determine the effect of a single dose of ketoconazole on the steady-state pharmacokinetic profile of JTK-853 and its metabolite M2 (one cohort only).

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) ≥18.0 kg/m2 and ≤30.0 kg/m2
2. Non-smokers or subjects who have stopped smoking at least 6 months prior to the Screening Visit
3. Female subjects must be either surgically sterile or postmenopausal

Exclusion Criteria:

1. History or presence of cardiac disease, including a family history of long-QT syndrome or unexplained sudden death
2. Have used any prescription medication, herbal product, or over-the-counter (OTC) medication (except acetaminophen) within four weeks prior to Day -1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 3 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of JTK-853 and metabolite M2 | 3 weeks
Time to reach peak or maximum concentration (tmax) for JTK-853 and metabolite M2 | 3 weeks
Area under the concentration-time curve during the dosing interval (AUCtau) for JTK-853 and metabolite M2 | 3 weeks
Elimination half-life associated with the terminal slope (λz) of a semilogarithmic concentration-time curve (t1/2) for JTK-853 and metabolite M2 | 3 weeks
Maximum concentration (Cmax) of JTK-853 and metabolite M2 after Ketoconazole administration | 3 weeks
Area under the concentration-time curve during the dosing interval (AUCtau) for JTK-853 and metabolite M2 after ketoconazole administration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Hoshino, D.V.M, Study Director — Akros Pharma Inc.
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States